CLINICAL TRIAL: NCT02872597
Title: A Phase I, Single Center, Placebo-Controlled, Blinded Pilot Study of Ipratropium Bromide in Children Admitted to the Intensive Care Unit With Status Asthmaticus
Brief Title: Phase I, Placebo-Controlled, Blinded Pilot Study of Ipratropium in Children Admitted to the ICU With Status Asthmaticus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Steven Shein, Attending Physician, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB #02-16-18
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Status Asthmaticus
MeSH Terms: conditions — Status Asthmaticus | interventions — Ipratropium; Albuterol, Ipratropium Drug Combination; Sodium Chloride; Saline Solution; Albuterol; Adrenal Cortex Hormones; Methylprednisolone; Prednisone; Dexamethasone; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): Inhaled ipratropium bromide 250mcg given via nebulization every 6 hours for up to 5 days
  Interventions: Drug: Ipratropium; Drug: Albuterol; Drug: corticosteroids
- Placebo (Placebo Comparator): Inhaled normal saline 1.25mL given via nebulization every 6 hours for up to 5 days
  Interventions: Drug: 0.9% Sodium Chloride; Drug: Albuterol; Drug: corticosteroids

INTERVENTIONS:
Drug: Ipratropium
  Other Names: Atrovent; Duoneb
  Arms: Treatment
Drug: 0.9% Sodium Chloride
  Other Names: Normal saline
  Arms: Placebo
Drug: Albuterol — albuterol prescribed by the clinical team per our PICU's "Asthma Carepath"
Drug: corticosteroids — systemic (IV or enteral) corticosteroid prescribed by the clinical team, typically methylprednisolone IV
  Other Names: methylprednisolone; prednisone; dexamethasone; prednisolone

SUMMARY:
This study is a Phase I study to investigate the addition of inhaled Ipratropium bromide to standard therapy in the treatment of severe asthma attacks in children admitted to the Pediatric Intensive Care Unit. Half of the subjects will receive inhaled Ipratropium, and half will receive an inhaled placebo.

DETAILED DESCRIPTION:
Status asthmaticus is an acute exacerbation of asthma that often requires treatment in a pediatric intensive care unit (PICU). Standard therapies for status asthmaticus include corticosteroids and bronchodilators, typically albuterol. Ipratropium bromide is also a bronchodilator, but has a different mechanism of action than albuterol. The addition of Ipraropium to children in the Emergency Room with severe asthma exacerbations improves outcomes, so many PICU doctors treat patients with status asthmaticus with Ipratropium. However, two studies of children hospitalized in the general wards of the hospital (not the PICU) show that the addition of Ipratropium to standard care does not effect clinical outcomes. This study is a first step towards determining in Ipratropium is helpful in PICU patients (like it is in ER patients) or if it not helpful (like it is in general ward patients).

ELIGIBILITY:
Inclusion Criteria:

* Admission to the PICU
* Treatment with continuous albuterol via the Asthma Carepath
* Enrollment occurred within 4 hours of starting continuous albuterol in the PICU
* Treatment with systemic corticosteroids by the clinical team

Exclusion Criteria:

* First episode of wheezing that prompted treatment with bronchodilators by medical personnel
* Prior enrollment in this study
* Patients with chronic lung disease requiring routine home oxygen use
* Allergy to inhaled ipratropium or inhaled saline
* Positive pressure ventilation (via an endotracheal tube or a non-invasive mask [e.g. CPAP (continuous positive airway pressure) or BiPAP])
* Pregnancy
* Tracheostomy
* Age < 2 years
* Age > 17 years
* Patient with pulmonary hypertension requiring daily therapy
* Patient with cyanotic congenital heart disease
* Cystic fibrosis

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2016-09-05 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-08-16 (Actual)

PRIMARY OUTCOMES:
Time to q2 Albuterol | typically 12-48 hours
  In our PICU, status asthmaticus patients are initially treated with continuous nebulization of albuterol. Per a standard assessment/scoring system, the patients are re-assessed each hour. When the patient's symptoms have sufficiently improved, the albuterol is weaned to 2.5mg given every 1hr ("q1hr albuterol") and, subsequently, to 2.5mg given every 2 hours ("q2hr Albuterol"). This outcome will measure the interval between the initiation of continuous albuterol and the second dose of q2hr Albuterol.

SECONDARY OUTCOMES:
PICU LOS (length of stay) | This outcome is assessed continually over the course of the study, typically 24-72 hours
  The time interval between admission to the PICU and discharge from the PICU, typically to the general ward. Patients are typically transferred to the general ward when they are receiving albuterol every 3 hours.
Hospital LOS (length of stay) | This outcome is assessed continually over the course of the study, typically 48-120 hours
  The time interval between admission to the hospital and discharge from the hospital. Patients are typically discharged from the hospital when they are receiving albuterol every 4 hours.

OTHER OUTCOMES:
Dry eyes | Adverse effects will be assessed 4-6hrs after each administration of study drug (and prior to the next administration of study drug)
  Report of dry eyes from the patient, their family or their clinical provider
Dry mouth | Adverse effects will be assessed 4-6hrs after each administration of study drug (and prior to the next administration of study drug)
  Report of dry mouth from the patient, their family or their clinical provider
Tremor | Adverse effects will be assessed 4-6hrs after each administration of study drug (and prior to the next administration of study drug)
  Report of tremor from the patient, their family or their clinical provider
Blurred vision | Adverse effects will be assessed 4-6hrs after each administration of study drug (and prior to the next administration of study drug)
  Report of blurred vision from the patient, their family or their clinical provider
Urinary retention | Adverse effects will be assessed 4-6hrs after each administration of study drug (and prior to the next administration of study drug)
  Report of urinary retention from the patient, their family or their clinical provider
Headache | Adverse effects will be assessed 4-6hrs after each administration of study drug (and prior to the next administration of study drug)
  Report of headache from the patient, their family or their clinical provider
Nausea/abdominal pain | Adverse effects will be assessed 4-6hrs after each administration of study drug (and prior to the next administration of study drug)
  Report of nausea/abdominal pain from the patient, their family or their clinical provider

CONTACTS AND LOCATIONS:
Locations (1):
- Rainbow Babies and Children's Hospital (of Univ. Hospitals Case Med. Center), Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Qureshi F, Pestian J, Davis P, Zaritsky A. Effect of nebulized ipratropium on the hospitalization rates of children with asthma. N Engl J Med. 1998 Oct 8;339(15):1030-5. doi: 10.1056/NEJM199810083391503. PMID 9761804
- [Background] Craven D, Kercsmar CM, Myers TR, O'riordan MA, Golonka G, Moore S. Ipratropium bromide plus nebulized albuterol for the treatment of hospitalized children with acute asthma. J Pediatr. 2001 Jan;138(1):51-58. doi: 10.1067/mpd.2001.110120. PMID 11148512
- [Background] Goggin N, Macarthur C, Parkin PC. Randomized trial of the addition of ipratropium bromide to albuterol and corticosteroid therapy in children hospitalized because of an acute asthma exacerbation. Arch Pediatr Adolesc Med. 2001 Dec;155(12):1329-34. doi: 10.1001/archpedi.155.12.1329. PMID 11732951
- [Background] Biagini Myers JM, Simmons JM, Kercsmar CM, Martin LJ, Pilipenko VV, Austin SR, Lindsey MA, Amalfitano KM, Guilbert TW, McCoy KS, Forbis SG, McBride JT, Ross KR, Vauthy PA, Khurana Hershey GK. Heterogeneity in asthma care in a statewide collaborative: the Ohio Pediatric Asthma Repository. Pediatrics. 2015 Feb;135(2):271-9. doi: 10.1542/peds.2014-2230. Epub 2015 Jan 19. PMID 25601985